CLINICAL TRIAL: NCT03160339
Title: A Phase 1 Two-Arm, Randomized, Double-blind, Active-controlled Study to Assess the Safety, Pharmacodynamics, and Immunogenicity of PXVX0047 (Adenovirus Type 4 and Type 7 Vaccine [A549 Cells], Live, Oral)
Brief Title: A Study to Assess the Safety, Pharmacodynamics, and Immunogenicity of PXVX0047
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PXVX-AD-047-001
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Adenoviral Infection
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PXVX0047 treatment group (Experimental): Subjects will receive PXVX0047 vaccine and Teva Placebo-to-Match
  Interventions: Biological: PXVX0047 Vaccine
- Teva Ad4/Ad7 treatment group (Active Comparator): Subjects will receive Teva Ad4/Ad7 vaccine and PXVX0047 Placebo-to-Match
  Interventions: Biological: Teva Ad4/Ad7 Vaccine

INTERVENTIONS:
Biological: PXVX0047 Vaccine — PXVX0047 is a live Adenovirus Type 4 (Ad4) / Adenovirus Type 7 (Ad7) vaccine for single-dose oral administration. The Ad4 and Ad7 strains in PXVX 0047 are unattenuated strains propagated in A549 human adenocarcinomic alveolar basal epithelial cells.
  Arms: PXVX0047 treatment group
Biological: Teva Ad4/Ad7 Vaccine — Teva Ad4/Ad7 is a live Adenovirus Type 4 (Ad4) / Adenovirus Type 7 (Ad7) vaccine for single-dose oral administration. The Ad4 and Ad7 strains in Teva Ad4/Ad7 are unattenuated strains propagated in WI-38 human diploid fibroblast cells.
  Arms: Teva Ad4/Ad7 treatment group

SUMMARY:
PXVX0047 (Adenovirus Type 4 and Type 7 Vaccine [A549 Cells], Live, Oral) is an investigational vaccine in development for the indication of active immunization against adenovirus infection. The primary goals of this Phase 1 study are to evaluate safety, pharmacodynamics (viral shedding), and immunogenicity of PXVX0047.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 to 35
* Seronegative for Ad4 and Ad7 by CPE-based assay
* (if female of childbearing potential) Using an acceptable method of contraception
* If male, subject agrees to use a highly effective method of contraception with female sexual partners of childbearing potential
* Able and willing to provide informed consent for study participation

Exclusion Criteria:

* Current acute febrile illness
* Current acute gastrointestinal illness
* Clinically significant cardiac, respiratory, or gastrointestinal disease
* (if female of childbearing potential) Pregnant or nursing, or who plan to become pregnant or nurse during the study
* Persons with occupations which may create an increased risk of transmission of vaccine virus (including but not limited to health care workers, child or elderly care providers, food handlers or preparers) who also have expected occupational contact with children less than 7 years of age, pregnant or nursing women, women of childbearing potential not using an acceptable method of contraception, or chronically ill or immunosuppressed individuals through Day 29.
* Expected household contact with children less than 7 years of age, pregnant or nursing women, women of childbearing potential not using an acceptable method of contraception, or chronically ill or immunosuppressed individuals through Day 29.
* Laboratory evidence of infection with Hepatitis B/C or HIV.
* History of severe allergic reaction (e.g. anaphylaxis) to any component of the vaccine.
* Inability to swallow capsules or tablets whole without chewing or crushing.
* Immunosuppressed individuals, including those treated or planned to be treated with systemic immunosuppressive medications within the 30 days prior to enrollment through 30 days after study treatment.
* Concomitant or planned use of other vaccines, investigational agents, cidofovir, ribavirin, or medications expected by the Investigator to have antiviral activity against adenovirus within 30 days prior to enrollment through Day 29.
* Any other condition that, in the opinion of the Investigator, creates an unacceptable risk to the subject.
* Any other condition that, in the opinion of the Investigator, may interfere with the conduct of the study or the validity of the data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of PXVX0047 by documenting the incidence of severity of solicited adverse events | From Day 1 through Day 15
  Incidence of severity of solicited adverse events include abdominal pain, nausea, vomiting, diarrhea, cough, nasal congestion, dyspnea, sore throat, headache, fever fatigue chills myalgia, arthralgia
Evaluate the safety and tolerability of PXVX0047 by documenting the incidence and severity of adverse events that are not solicited. | From Day 1 through Day 29
  Unsolicited adverse events include clinical significant laboratory abnormalities
Evaluate the induction of anti-Ad4 neutralizing activity by measuring the Ad4 and Ad7 seroconversion rate | From Day 1 to Day 29
  The Ad4 seroconversion rate is defined as the percent of subjects seroconverted (i.e. with a 4-fold or greater rise over baseline in neutralizing antibody titer) to Ad4 as determined by cytopathic-effect (CPE)-based assay
Evaluate the induction of anti-Ad7 neutralizing activity by measuring the Ad7 seroconversion rate | From Day 1 to Day 29
  The Ad7 seroconversion rate is defined as the percent of subjects seroconverted (i.e. with a 4-fold or greater rise over baseline in neutralizing antibody titer) to Ad7 as determined by cytopathic-effect (CPE)-based assay

SECONDARY OUTCOMES:
Evaluate the pharmacodynamics of PXVX0047 by measuring the shedding of Ad4 viruses via the GI tract | Days 4, 8, 15, 22, and 29
  Shedding of Ad4 via the GI tract, as assessed by rectal swabs
Evaluate the pharmacodynamics of PXVX0047 by measuring the shedding of Ad7 viruses via the GI tract | Days 4, 8, 15, 22, and 29
  Shedding of Ad7 via the GI tract, as assessed by rectal swabs
Evaluate the pharmacodynamics of PXVX0047 by measuring the shedding of Ad4 viruses via the respiratory tract | Days 4, 8, 15, 22, and 29
  Shedding of Ad4 via the respiratory tract, as assessed by throat swabs.
Evaluate the pharmacodynamics of PXVX0047 by measuring the shedding of Ad7 viruses via the respiratory tract | Days 4, 8, 15, 22, and 29
  Shedding of Ad7 via the respiratory tract, as assessed by throat swabs.
Evaluate the pharmacodynamics of PXVX0047 by measuring the presence of Ad4 viremia | Days 4, 8, 15, 22, and 29
  Presence of Ad4 viremia in the blood
Evaluate the pharmacodynamics of PXVX0047 by measuring the presence of Ad7 viremia | Days 4, 8, 15, 22, and 29
  Presence of Ad7 viremia in the blood
Evaluate the immunogenicity of PXVX0047 by measuring Ad4 seroconversion rates | Through Day 57
  The Ad4 seroconversion rates, measured independently, determined by luciferase and CPE-based assays
Evaluate the immunogenicity of PXVX0047 by measuring Ad7 seroconversion rates | Through Day 57
  The Ad7 seroconversion rates, measured independently, determined by luciferase and CPE-based assays
Evaluate the immunogenicity of PXVX0047 by measuring cumulative Ad4 seroconversion rates | Through Day 57
  The cumulative Ad4 seroconversion rates, measured independently, where cumulative seroconversion through a particular visit is defined as having seroconverted at or prior to that visit.
Evaluate the immunogenicity of PXVX0047 by measuring cumulative Ad7 seroconversion rates | Through Day 57
  The cumulative Ad7 seroconversion rates, measured independently, where cumulative seroconversion through a particular visit is defined as having seroconverted at or prior to that visit.
Evaluate the immunogenicity of PXVX0047 by measuring geometric mean titer | Through Day 57
  The geometric mean titer (GMT) of neutralizing antibodies to Ad4, measured independently
Evaluate the immunogenicity of PXVX0047 by measuring geometric mean titer | Through Day 57
  The geometric mean titer (GMT) of neutralizing antibodies to Ad7, measured independently
Evaluate the immunogenicity of PXVX0047 by measuring the fold-rise over baseline of neutralizing antibodies to Ad4 viruses | Through Day 57
  The fold-rise over baseline in neutralizing antibodies to Ad4, measured independently
Evaluate the immunogenicity of PXVX0047 by measuring the fold-rise over baseline of neutralizing antibodies to Ad7 viruses | Through Day 57
  The fold-rise over baseline in neutralizing antibodies to Ad7, measured independently
Evaluate the immunogenicity of PXVX0047 by measuring the cellular immune responses to Ad4 viruses | At Days 29 and 57.
  The cellular immune responses to Ad4, measured independently
Evaluate the immunogenicity of PXVX0047 by measuring the cellular immune responses to Ad7 viruses | At Days 29 and 57.
  The cellular immune responses to Ad7, measured independently

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beaty S, Collins N, Karasavvas N, Kuschner R, Hang J, Adhikari A, Maljkovic Berry I, Fung C, Walls S, Betancourt E, Mendy J, Lock M, Gierman E, Bennett S, Shabram P, Warfield K. A Phase 1 Two-Arm, Randomized, Double-Blind, Active-Controlled Study of Live, Oral Plasmid-Derived Adenovirus Type 4 and Type 7 Vaccines in Seronegative Adults. Vaccines (Basel). 2023 Jun 12;11(6):1091. doi: 10.3390/vaccines11061091. PMID 37376480